CLINICAL TRIAL: NCT02917187
Title: An Exploratory, Randomized, Double-Blind, Crossover Study to Compare the Efficacy and Safety of BIIB074 Versus Placebo in the Treatment of Primary Inherited Erythromelalgia
Brief Title: A Phase 2a Study of BIIB074 in the Treatment of Erythromelalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1014802-205
Record Dates: First submitted 2016-07-19; First posted 2016-09-28 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Primary Inherited Erythromelalgia
MeSH Terms: interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized Group 1 (Experimental): After two week run-in, BIIB074 three times a day (TID) followed by placebo (TID) after two week washout period
  Interventions: Drug: BIIB074; Drug: Placebo
- Randomized Group 2 (Experimental): After two week run-in, Placebo three times a day (TID) followed by BIIB074 (TID) after two week washout period
  Interventions: Drug: BIIB074; Drug: Placebo

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm
  Other Names: CNV1014802
Drug: Placebo — Matched placebo

SUMMARY:
The primary objective of the study is to investigate the efficacy of repeat oral dosing of BIIB074 on paroxysmal pain in participants with Primary Inherited Erythromelalgia (EM). The secondary objective of the study is to investigate the efficacy of repeat oral dosing of BIIB074 on varying additional aspects of pain in participants with EM; and to investigate the safety and tolerability of repeat oral dosing of BIIB074 in participants with EM.

DETAILED DESCRIPTION:
This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of primary inherited EM with family history of EM made at least 3 months from initial diagnosis.
* Failed at least one prior treatment for EM (defined as an inadequate response or intolerance to treatment).
* Approved concomitant medications must have been stable for at least 4 weeks prior to day 1.

Key Exclusion Criteria:

* Positive screening Hepatitis B surface antigen or positive Hepatitis C antibody result.
* Received nerve blocks and/or steroid injections for neuropathic pain within 4 weeks prior to Day 1.
* Males whose partner is pregnant.
* Failed at least one prior treatment for EM (defined as an inadequate response or intolerance to treatment).

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Weekly average severity of paroxysms | Day 1 to Week 12
  11-point Pain Intensity Numerical Rating Scale (PI-NRS) is used to assess EM paroxysmal pain. PI-NRS is an 11-point pain intensity numerical rating scale, where 0=no pain and 10=worst possible pain.
  Weekly average is defined as the total of severity scores during a week divided by the total number of paroxysms during that week.

SECONDARY OUTCOMES:
Weekly maximum severity of paroxysms | Day 1 to Week 12
  The weekly maximum severity is the maximum paroxysm severity recorded by a participant in a given week.
Weekly average and maximum number of paroxysms | Day 1 to Week 12
Weekly average and weekly maximum duration of paroxysms | Day 1 to Week 12
Weekly average and weekly maximum of daily background pain | Day 1 to Week 12
  Each participant provides a daily background pain score via a diary that records background daily pain intensity using a numerical rating scale from 0-10 with higher scores indicating worse pain.
Patient Global Impression of Change (PGIC) score | Day 1 to Week 12
  PGIC is a 7-point self-report scale depicting a participant's rating of overall improvement. Participants rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Weekly average and weekly maximum number of pain-mitigating activities | Day 1 to Week 12
  Participant diary is used to record pain mitigating cooling activities that include but are not limited to use of cold water or fan.
Weekly average and weekly maximum duration of pain-mitigating activities | Day 1 to Week 12
  Participant diary is used to record pain mitigating activities that include but are not limited to use of cooling, and breathing/relaxation and mental imagery techniques.
Use of rescue medication | Day 1 to Week 13
Weekly average and weekly maximum of the daily sleep interference scale | Day 1 to Week 12
  Daily Sleep Interference Scale (DSIS) describes how much EM pain interfered with the participant's sleep with 0 indicating "pain did not interfere with sleep" and 10 indicating "pain completely interfered with sleep".
Weekly average and weekly maximum number of awakenings at night due to EM pain | Day 1 to Week 12
Number of participants experiencing adverse events (AEs) and serious adverse events (SAEs) | Up to Week 13
Number of participants with clinically significant vital sign abnormalities | Up to Week 13
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to Week 13
Number of participants with clinically significant laboratory safety test abnormalities | Up to Week 13
Columbia-Suicide Severity Rating Scale (C-SSRS) assessment | Up to Week 13
  C-SSRS is a suicidal ideation rating used to evaluate suicidality. It rates an individual's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent."

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- United States (5):
  - Research Site, Birmingham, Alabama
  - Research SIte, New London, Connecticut
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Plano, Texas
  - Research Site, Morgantown, West Virginia